CLINICAL TRIAL: NCT06604793
Title: Effects of Equal-volume Creatine Supplementation With Different Dosing Strategies on Body Composition and Muscle Performance in Young Healthy Adults
Brief Title: Creatine Supplementation in Young Healthy Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Iovate Health Sciences International Inc (Industry)
Responsible Party: Principal Investigator, Darren Candow, Professor, University of Regina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 834
Record Dates: First submitted 2024-09-17; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Improve Muscle Performance in Young Adults
MeSH Terms: interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Creatine Bolus (Experimental): (Serving 1: 5 grams of creatine monohydrate + 3 grams of placebo in the morning; Serving 2: 8 grams of placebo in the evening) for 21 days.
  Interventions: Dietary Supplement: Creatine
- Creatine Intermittent (Experimental): (Serving 1: 2.5 grams of creatine monohydrate + 5.5 grams of placebo in the morning; Serving 2: 2.5 grams of creatine monohydrate + 5.5 grams of placebo in the evening) for 21 days.
  Interventions: Dietary Supplement: Creatine
- Placebo (Placebo Comparator): (Servings 1: 8 grams of placebo in the morning; Serving 2: 8 grams of placebo in the evening) for 21 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Creatine — Creatine monohydrate
  Arms: Creatine Bolus; Creatine Intermittent
Dietary Supplement: Placebo — Maltodextrin
  Arms: Placebo

SUMMARY:
The purpose is to compare the effects of bolus ingestion (5 grams) vs. intermittent ingestion (2 x 2.5 grams) of creatine supplementation vs. placebo for 21 days on measures of body composition (lean tissue mass-indicator of muscle mass, total body water) and muscle performance (i.e., power, strength, endurance).

DETAILED DESCRIPTION:
Creatine is a naturally occurring compound produced in the liver and brain. Creatine can also be found in food products such as red meat and seafood or through commercially available manufactured creatine products (i.e. creatine supplementation).

Evidence-based research shows that creatine supplementation improves measures of body composition and muscle performance. However, the optimal creatine supplementation protocol to achieve these benefits is unknown.

ELIGIBILITY:
Inclusion Criteria:

* if you are 18-39 years of age
* if you have not been performing resistance training for at least 4 weeks prior to the start of the study.

Exclusion Criteria:

* if you are pregnant or nursing
* have taken creatine monohydrate within 30 days prior to the start of the study
* if you have pre-existing allergies to the placebo (corn-starch maltodextrin)

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Whole-body lean mass (kg) | baseline, day 21
  Bioelectrical impedance analysis
Strength | baseline, day 21
  1-repetition maximum leg press and chest press (kg)
Endurance | baseline, day 21
  Repetitions to fatigue for leg press and chest press (total number)
Hydration | baseline, day 21
  Total body water (kg) using bioelectrical impedance analysis
Power | baseline, day 21
  Vertical Jump (cm)
Power | baseline, day 21
  Medicine Ball Throw (feet)

CONTACTS AND LOCATIONS:
Overall Officials: Darren Candow, Principal Investigator — University of Regina
Locations (1):
- University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No